CLINICAL TRIAL: NCT00792675
Title: Evaluation of the Effect of Exercise on Disease Activity and Immune Parameters in Persons With Rheumatoid Arthritis
Brief Title: Effect of Exercise on the Disease Activity of Rheumatoid Arthritis
Acronym: RA&Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Arthritis Foundation (Other); Nebraska Chapter Arthritis Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0267-02-FB
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
Keywords: exercise; disease activity; inflammation; resistance training; rehabilitation
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Exercise consists of 30 minutes of treadmill exercise at approximately 85% of heart rate max and 2 sets of 6 resistance weight lifting exercises resulting in volitional fatigue at 12 to 15 repetitions.
  Interventions: Other: Aerobic and resistance exercise training

INTERVENTIONS:
Other: Aerobic and resistance exercise training — Exercise was performed 3 times per week. It consisted of 30 minutes of treadmill exercise at approximately 85% of heartrate max and 2 sets of 6 resistance weight lifting exercises resulting in volitional fatigue at 12 to 15 repetitions.

SUMMARY:
This study will evaluate the effect of exercise on the number of swollen and tender joints associated with rheumatoid arthritis after a 12 week exercise program of treadmill walking and weightlifting.

DETAILED DESCRIPTION:
The goal of this study was to evaluate the effect of exercise on the number of swollen and tender joints associated with rheumatoid arthritis. It was hypothesized that persons would have less inflammation associated with rheumatoid arthritis after a 12 week exercise program of treadmill walking and weighlifting. Immune parameters were measured to determine potential mechanisms responsible for changes in inflammation with exercise.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of RA according to the ACR 1989 Criteria at least 6 months prior to enrollment in the study, but not longer than 12 years
* age 19 to 65 years old
* stable regimen of medication for 2 months with less than 10 mg/day of oral corticosteroids
* currently exercise < 2x/week for less than 30 minutes at less than 60% of his/her age predicted maximum heart rate
* Subjects must pass the Physical Activity Readiness Scale Questionnaire (PAR-Q)

Exclusion Criteria:

* other serious health problems
* intra-articular injection within 6 weeks
* total joint replacement of the large joints
* use of beta-blockers
* inability to complete the submaximal exercise test

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2006-04-01 (Actual); Study Completion 2006-11-01 (Actual)

PRIMARY OUTCOMES:
Swollen Joint Count | 12 Weeks
Tender Joint Count | 12 Weeks

SECONDARY OUTCOMES:
Pain (visual Analog Scale) | 12 Weeks
Modified-Health Assessment Questionnaire | 12 Weeks
Estimated Aerobic Capacity (VO2max) | 12 weeks
SF-36 | 12 Weeks
Patient Global Assessment | 12 Weeks
Practitioner Global Assessment | 12 Weeks
Timed-Stands Test | 12 Weeks
50 Foot Walk Test | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Bilek, PhD, PT, Principal Investigator — University of Nebraska
Locations (1):
- Physical Activity Lab, University of Nebraska Omaha, Omaha, Nebraska, United States